CLINICAL TRIAL: NCT02478866
Title: Safety and Pharmacokinetics of BPI-9016M in Patients With Advanced Solid Tumors: A Phase Ia Study, Open-label, Dose-escalation Study
Brief Title: Safety and Pharmacokinetics of BPI-9016M in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-CM-I01
Record Dates: First submitted 2015-05-21; First posted 2015-06-23 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2017-04

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BPI-9016M (Experimental): Seven dose cohorts will be evaluated, including 100mg, 200mg, 300mg, 450mg, 600mg, 800mg, 1000mg. BPI-9016M will be administered orally to patients once daily for each dose cohort.
  Interventions: Drug: BPI-9016M

INTERVENTIONS:
Drug: BPI-9016M — Seven dose cohorts will be evaluated, including 100mg, 200mg, 300mg, 450mg，600mg, 800mg, 1000mg. BPI-9016M will be administered orally to patients once daily for each dose cohort.
  Other Names: No other name currently

SUMMARY:
BPI-9016M is a novel, highly potent and selective small-molecule inhibitor of c-Met/Axl kinase. In preclinical studies, it demonstrated strong activity in vitro and in vivo against c-Met/Axl kinase and its downstream signaling targets, and inhibited tumor cell growth. This first-in-human study is conducted to assess the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT), to evaluate the pharmacokinetics, safety and preliminary anti-tumor activity of BPI-9016M with single doses and multiple doses.

DETAILED DESCRIPTION:
This is a phase Ia study, first-in-human, open-label, dose-escalation study of BPI-9016M administered orally once daily (QD) to patients with locally advanced or metastatic solid tumors.The study is designed to evaluate the safety, tolerability, and pharmacokinetics of single dose and multiple doses of BPI-9016M.

All patients will be followed up for adverse events during the study treatment and 28 days after the last dose of study drug. Subjects of this study will be permitted to continue therapy only when BPI-9016M is well tolerated, and tumor response or stable disease is seen.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, locally advanced, or metastatic solid tumor that progressed, or failed to respond to, at least one prior systemic therapy
* Evaluable or measurable disease per Response Evaluation Criteria in Solid Tumors(RECIST1.1)
* Life expectancy ≥3 months
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Adequate bone marrow, hepatic, and renal function
* Patients of child bearing potential must agree to take contraception during the study and for 90 days after the last day of treatment
* Signed Informed Consent Form

Exclusion Criteria:

* Prior treatment with agents of HGF/c-Met inhibitors or HGF/c-Met antibody(Including Crizotinib,Cabozantinib,Volitinib etc.)
* Any anti-cancer therapy, including chemotherapy, hormonal therapy, biologic therapy or radiotherapy within 4 weeks prior to initiation of study treatment
* History of organ transplant; had surgery or severe injury within 4 weeks
* Adverse events from prior anti-cancer therapy that have not resolved to Grade ≤ 2, except for alopecia
* Any evidence of severe or uncontrolled systemic diseases, including CTCAE 3 or higher active infection, unstable angina pectoris, congestive cardiac failure and severe liver/renal or metabolic disease
* Pregnant (positive pregnancy test) or lactating women
* Inability to take oral medication, prior surgical procedures affecting absorption, or active peptic ulcer disease
* Brain/meninges metastases unless asymptomatic, stable and not requiring steroids for maintenance
* Active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV)
* Inability to comply with study and follow-up procedures
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the patient at high risk from treatment complications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-08-11 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Participants with Adverse Events | 24 months
  The safety and tolerability variables include adverse events, physical examinations, vital signs (specifically including blood pressure), clinical laboratory evaluations including serum chemistry, hematology(Maximum Tolerated Dose) , and urinalysis (with detailed sediment analysis, proteinuria, and 24-hour urine for collection for protein), and electrocardiograms (ECGs) in triplicate,Incidence and nature of DLTs(Dose-Limiting Toxicity),To determine the MTD (Maximum Tolerated Dose).

SECONDARY OUTCOMES:
Cmax | 1 month
  Day 1-3 for single dose, and day 1-21 for steady state
Half-life time | 1 month
  Day 1-3 for single dose, and day 1-21 for steady state
Tmax | 1 month
  Time to Cmax

OTHER OUTCOMES:
Progression-free survival | 18-24 months

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, MD, Study Chair — Department of Medical Oncology, Cancer Institute/Hospital, Chinese Academy of Medical Sciences; Pei Hu, MD, Study Chair — Peking Union Medical College Hospital
Locations (2):
- China (2):
  - Department of Medical Oncology, Cancer Institute/Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking Union College Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu X, Zheng X, Yang S, Wang L, Hao X, Cui X, Ding L, Mao L, Hu P, Shi Y. First-in-human phase I study of BPI-9016M, a dual MET/Axl inhibitor, in patients with non-small cell lung cancer. J Hematol Oncol. 2020 Jan 16;13(1):6. doi: 10.1186/s13045-019-0834-2. PMID 31948451